CLINICAL TRIAL: NCT05270785
Title: Preventing Suicide Among Sexual and Gender Diverse Young Adults in Primary Care in Texas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible participants during study time period
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth Arnold, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0351; SP-2020C3-210 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Suicidal Ideation
Keywords: suicidal ideation; depression; suicide; sexual and gender minority youth
MeSH Terms: conditions — Suicidal Ideation; Depression; Suicide; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suicidal Teens Accessing Treatment - Primary Care (STAT-PC) (Experimental): This group will undergo a brief, suicide prevention intervention based on motivational interviewing that focuses on mental health care seeking behavior, problem-solving, and referrals plus brief case management
  Interventions: Other: STAT-PC
- Youth-Nominated Support Team (YST-III) (Experimental): This group will undergo a brief, suicide prevention intervention originally developed for youth who have been psychiatrically hospitalized due to a suicide attempt or suicidal ideation that has been adapted
  Interventions: Other: YST-III

INTERVENTIONS:
Other: STAT-PC — STAT-PC is an adapted version of Suicidal Teens Accessing Treatment after an ED Visit (STAT-ED). It is a brief intervention based on motivational interviewing (MI) that focuses on mental health care seeking behavior, problem-solving, and referrals plus brief case management (2-3 follow-up calls). The intervention will consist of an initial session with the youth focusing on accessing mental health care plus two case management calls. The interventionist will also be available to assist with referrals for connection to other services later during the study period as needed for up to two months. The intervention may include contact with the youth's mental health provider to make sure linkages are made.
  Arms: Suicidal Teens Accessing Treatment - Primary Care (STAT-PC)
Other: YST-III — YST-III is an adapted version of Youth-Nominated Support Team for Suicidal Adolescents (YST-II). The intervention is a brief intervention developed for youth who have been psychiatrically hospitalized due to a suicide attempt or suicidal ideation (SI). Participants will nominate 1-2 supportive adults (age 18 and older) from their lives who agree to provide ongoing contact and support for up to 2 months. YST-III will include an introductory session with the youth who will nominate their support persons plus referrals for mental health services. The support persons will receive training on how to best support their youth partner and then ongoing calls to support them in working with their youth partner for up to 2 months.
  Arms: Youth-Nominated Support Team (YST-III)

SUMMARY:
The aim of this pilot study is to reduce suicide among sexual and gender diverse youth ages 18-24 years old. This pilot study will compare two brief suicide prevention interventions that have been adapted for use with this population to use in primary care via telehealth and will recruit 40 youth from 4-6 primary care clinics in the Dallas and Austin, Texas metropolitan areas. Each clinic will be randomly assigned to deliver one of the two study interventions.

DETAILED DESCRIPTION:
This is a cluster randomized study focused on youth suicide prevention which will recruit 40 youth from four primary care clinics serving sexual and gender diverse young adults in the Dallas and Austin, TX metropolitan areas. Each clinic will recruit 10 youth. Two clinics will be randomly assigned to deliver each of the two study interventions. The interventions are adapted versions of two existing, brief suicide prevention interventions: 1) Suicidal Teens Accessing Treatment after an ED Visit (STAT-ED) is a brief intervention based on motivational interviewing that focuses on mental health care seeking behavior, problem-solving, and referrals plus brief case management; and 2) Youth-Nominated Support Team for Suicidal Adolescents (YST-II) is a brief intervention developed for youth who have been psychiatrically hospitalized due to a suicide attempt or suicidal ideation. The revised interventions will be called STAT-PC and YST-III. For YST III, participants will identify 1-2 supportive adults from their lives who agree to provide ongoing contact and support. The interventions will last two months. Primary and secondary outcome assessments will be done at baseline and/or at 2 months.

To be eligible, participants must report risk factors for suicide based on screening questions that will be implemented in our primary clinic sites.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18-24 at the time of enrollment; and
* not have received mental health services in the past 90 days, excluding medication;
* English-speaking, and
* screen positive for suicidal ideation.

Exclusion Criteria:

* are actively suicidal
* have a developmental disability that would preclude them from participating in the study intervention or
* who are impaired due to psychosis, mania, or substance use that would prevent them from providing consent.
* Participants will also be excluded at YST-III sites if they are unable to identify a minimum of one support person to participate in the intervention with them.

Those who are excluded will be provided with referrals for treatment services.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — To enroll, participants must identify as a sexual or gender minority individual (i.e., LGBTQ+) and be a patient of the one the clinic sites
Enrollment: 3 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change in suicidal ideation as measured by ASIQ | Baseline, 2 months
  Change in suicidal ideation is measured by Adult Suicidal Ideation Questionnaire (ASIQ). It is a 25-item, self-report assessment of suicidal thoughts designed specifically for adult populations. Possible scores range from 1 (Not at All) to 6 (Extreme), with lower scores indicating less severe suicidal ideation (better outcome)

SECONDARY OUTCOMES:
Change in number of mental healthcare service utilization as measured by ED-STARS mental health service utilization check list | Baseline, 2 months
  Change in number of mental healthcare service utilization is measured by Emergency Department Screen for Teens at Risk for Suicide (ED-STARS) mental health service utilization check list which will be used to assess the number of different types of mental health services that participants receive including inpatient psychiatric services, emergency department visits, medication management, and psychotherapy/counseling.
Number of past 2 months suicide attempts at baseline | Baseline
  Past 2 months suicide attempts is measured by suicide attempt question from the Columbia-Suicide Severity Rating Scale (CSSRS) which will assess the number of suicide attempts.
Number of lifetime suicide attempts at baseline | Baseline
  Suicide attempts is measured by suicide attempt question from the Columbia-Suicide Severity Rating Scale (CSSRS) which will assess the number of suicide attempts.
Number of suicide attempts at 2 months | 2 months
  Suicide attempts is measured by suicide attempt questions from the Columbia-Suicide Severity Rating Scale (CSSRS) which will assess the number of suicide attempts.
Change in depressive symptoms as measured by CESD-R | Baseline, 2 months
  Change in depressive symptoms is measured by Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) which is a 20-item measure of depression that assesses the duration symptoms across a period of two weeks. Possible scores range from 0-60, with lower scores indicating less depressive symptoms (better outcome).
Change in social support as measured by MSPSS | Baseline, 2 months
  Change in social support is measured by Multidimensional Scale of Perceived Social Support (MSPSS) which is a 12-item measure with three subscales that assesses family, friend, and significant other support. Response categories are on a 7-point Likert-scale from 1=very strongly disagree to 7=very strongly agree. The overall score will be used to assess change. The 12-item MSPSS scale has a mean continuous score ranging from 1-84. Higher scores indicate greater perceived social support (better outcome).
Change in internalized stigma as measured by ITS-adapted | Baseline, 2 months
  Change in internalized stigma is measured by Internalized Transphobia Scale (ITS) - adapted. Internalized stigma will be measured by an adapted version of the Internalized Transphobia Scale (ITS). The measure consists of 22 questions. Possible score ranges from 1-4 with lower scores indicating less internalized stigma (better outcome)
Number of deaths by suicide at 2 months | 2 months
  The data on any reported deaths due to suicide during the study period will be collected.

OTHER OUTCOMES:
Number of participants who had access to means for suicide at baseline | Baseline
  This is a descriptive measure with patient reported Yes/ No responses and if yes, to categorize the means for suicide.
Number of participants who had access to means for suicide at 2 months | 2 months
  This is a descriptive measure with patient reported Yes/ No responses and if yes, to categorize the means for suicide.
Proportion of participants who screened and met criteria | Last day of study recruitment period (approx. week 14)
  Proportion of participants who screened and met criteria is obtained at the last day of the study recruitment period.
Proportion of participants who enrolled in the study | Last day of study recruitment period (approx. week 14)
  Proportion of participants who enrolled in the study is obtained at the last day of the study recruitment period.
Number of participants who decide not to participate | 2 months post-intervention
  For potential study candidates who decide not to participate, refusal reason will be logged.
Intervention acceptability | 1 month post-intervention
  Intervention acceptability will be measured by asking participants to rate the extent to which they agree with 4 statements about the study intervention received on a scale of 1 to 4 where 1 is strongly disagree and 4 is strongly agree
Study feasibility | 1 month post-intervention
  Study feasibility will be measured by asking participants to rate the extent to which they agree with 5 statements about the study on a scale of 1 to 4 where 1 is strongly disagree and 4 is strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Arnold, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No